CLINICAL TRIAL: NCT02711267
Title: An Exploratory Study to Evaluate Dermal Open Flow Microperfusion's (dOFM) Ability to Assess Bioequivalence and Non-bioequivalence of Topical Acyclovir Formulations in Healthy Volunteers
Brief Title: Bioequivalence of Topical Acyclovir in Healthy Volunteers
Acronym: FDA_BE1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Collaborators: Joanneum Research Forschungsgesellschaft mbH (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: FDA_BE1
Record Dates: First submitted 2015-07-29; First posted 2016-03-17 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Dermatologic Disorders
Keywords: Open Flow Microperfusion
MeSH Terms: conditions — Skin Diseases | interventions — Acyclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Phase 1: Optimization Study (Experimental): 6 subjects will be included in this study, each with 3 application sites on the arm and 3 on the leg. 2 dOFM probes (OFM Probe) will be implanted per site resulting in 12 dOFM probes per subject (operated by OFM pump). On each the arm and the leg the proximal and distal site of the 3 adjacent sites will be treated by 5% Zovirax® cream. The central site on arm and leg will be left untreated in order to test a potential lateral carry-over of acyclovir from one application site to the other. Blood samples will be taken to test for uptake into the blood stream and redistribution to other application sites.
  Interventions: Drug: 5% Zovirax® cream; Procedure: OFM; Device: OFM Probe; Device: OFM Pump
- Phase 2: Formulation Study (Experimental): 6 subjects will be included in this study, each with 3 application sites on the arm and 3 on the leg. 2 dOFM probes will be implanted per site resulting in 12 dOFM probes per subject. Different topical 5% acyclovir formulations currently available on the market will be tested. One application site on the arm and one on the leg will be used for U.S. Zovirax® cream 5% application. The remaining two application sites on the arm and the remaining 2 on the leg will be used to randomly administer two of the remaining formulations (5% Aciclostad cream, 5% Aciclovir cream 1A Pharma, 5% Zovirax® cream (Austria), 5% Zovirax Cold Sore Cream) according to an application pattern.
  Interventions: Drug: 5% Zovirax® cream; Drug: 5% Aciclostad cream; Drug: 5% Aciclovir cream 1A Pharma; Drug: 5% Zovirax Cold Sore Cream; Drug: 5% Zovirax® cream (Austria); Procedure: OFM; Device: OFM Probe; Device: OFM Pump
- Phase 3: Pilot BE study (Experimental): 4 subjects will be included in the pilot BE study with 3 application sites on each leg. 2 dOFM probes will be implanted per site resulting in 12 dOFM probes per subject. One reference drug product (R) and one test drug product (T) will be applied on the application sites in order to test for BE between duplicate sites with R applied, and to test for non-BE between application sites with R and T applied.
  Interventions: Drug: 5% Zovirax® cream; Drug: 5% Aciclovir cream 1A Pharma; Procedure: OFM; Device: OFM Probe; Device: OFM Pump
- Phase 4: Main BE Study (Experimental): 20 subjects will be included in the pilot BE study with 3 application sites on each leg. 2 dOFM probes will be implanted per site resulting in 12 dOFM probes per subject. One reference drug (R) and one test drug (T) will be applied on the application sites in order to test for BE between duplicate sites with R applied and to test for non-BE between application sites with R and T applied.
  Interventions: Drug: 5% Zovirax® cream; Drug: 5% Aciclovir cream 1A Pharma; Procedure: OFM; Device: OFM Probe; Device: OFM Pump

INTERVENTIONS:
Drug: 5% Zovirax® cream — (manufactured by GlaxoSmithKline Pharma in Canada, distributed in the USA by Valeant Pharmaceuticals North America LCC, Bridgewater,NJ 08807)
  Other Names: Aciclovir
Drug: 5% Aciclostad cream — (STADA Arzneimittel GmbH, Vienna, Austria)
  Other Names: Aciclovir
  Arms: Phase 2: Formulation Study
Drug: 5% Aciclovir cream 1A Pharma — (1A Pharma GmbH, Vienna, Austria)
  Other Names: Aciclovir
  Arms: Phase 2: Formulation Study; Phase 3: Pilot BE study; Phase 4: Main BE Study
Drug: 5% Zovirax Cold Sore Cream — (GlaxoSmithKline Consumer Health Care, Brendfort, UK; Marketing authorization holder: Beeham Group PLC, Brendfort, UK)
  Other Names: Aciclovir
  Arms: Phase 2: Formulation Study
Drug: 5% Zovirax® cream (Austria) — (GlaxoSmithKline Pharma GmbH, Vienna, Austria)
  Other Names: Aciclovir
  Arms: Phase 2: Formulation Study
Procedure: OFM — Sampling method for interstitial fluid
  Other Names: Open Flow Microperfusion
Device: OFM Probe — Sampling probe used during OFM
  Other Names: 'DEA15003' (linear type, 0.5mm OD, 15mm open mesh)
Device: OFM Pump — Pump used to operate OFM probes
  Other Names: 'MPP102' (wearable, operates 3 to 6 probes)

SUMMARY:
The overall aim of this clinical study is to investigate the ability of dermal open flow microperfusion to assess bioequivalence and non-bioequivalence of acyclovir formulations in the skin of healthy volunteers.

DETAILED DESCRIPTION:
This will be a single center, open label, exploratory research study to evaluate the BE of already marketed formulations of acyclovir in dermal interstitial fluid (ISF) in healthy volunteers using dOFM. The study will be conducted at the Clinical Research Center at the Medical University Graz. dOFM represents the most reliable way to sample interstitial fluid from skin, since it provides diluted but otherwise unchanged dermal interstitial fluid. To assess BE and non-BE, we have designed the experiments in such a way that each subject can serve as its own control. Each subject will have two sets of BE and non-BE pairs in parallel. This study is designed to test dOFM, a new sampling method that allows measurement of skin penetration. Measurement of skin penetration enables the reduction of the impact of inter-subject variability and therefore decreases the number of subjects needed to achieve statistical significance.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained before any assessment is performed.
2. Male and female subjects 21 to 50 years of age inclusive and in good health as determined by past medical history, physical examination, vital signs, electrocardiogram, and laboratory tests at screening.
3. Able to communicate well with the investigator, to understand and comply with the requirements of the study.

Exclusion Criteria:

1. Use of other investigational drugs at the time of enrollment, or within 30 days or 5 half-lives of enrollment, whichever is longer; or longer if required by local regulations, and for any other limitation of participation in an investigational trial based on local regulations.
2. History of hypersensitivity to any of the study drugs or to drugs of similar chemical classes.
3. Use of topical corticosteroids or systemic immunosuppression within the last 3 weeks (for topicals) or 3 months (systemic medication)
4. A history of clinically significant ECG abnormalities, or any of the following ECG abnormalities at screening or baseline.

   * PR > 220 msec
   * QRS complex > 120 msec
   * Long QT syndrome
   * QTcF > 430 msec males, > 450 females
5. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG (human chorionic gonadotropin) laboratory test (> 10 mIU/mL).
6. Significant medical problems, including but not limited to the following: uncontrolled hypertension (≥160 systolic /95 diastolic mm Hg), congestive heart failure [New York Heart Association status of class III or IV].
7. Screening total WBC count <3,500cells/µL, or platelets <140,000cells/µL or neutrophils <2,000cells/µL or hemoglobin <12 g/dL / <13.5g/dL for female / male.
8. Active systemic infections during the last two weeks (exception: common cold) prior to enrollment.
9. A febrile illness within 72 hours, or major dental work within 8 days, prior to first dosing.
10. History of immunodeficiency diseases, including a positive HIV (ELISA and Western blot) test result.
11. A positive Hepatitis B surface antigen (HBsAg) or Hepatitis C test result.
12. Inability or unwillingness to undergo repeated catheterization and / or venipuncture (e.g., because of poor tolerability or lack of access to veins). Inability or unwillingness of having a skin biopsy if consent was given.
13. Any medical or psychiatric condition or clinical laboratory abnormalities which, in the Investigator's opinion, would interfere with interpretation of study results and/or make the participant likely not to adhere to the protocol or complete the study per protocol.
14. History of venous thrombosis or known genetic predisposition to thromboembolic events
15. Subjects prone to keloid or hypertrophic scar formation or any wound healing disorder as visible by checking the vaccine insertion points on upper arm.
16. Fear of needles (belonephobia)
17. Recent (within the last three [3] years) and/or recurrent history of autonomic dysfunction (e.g., recurrent episodes of fainting, palpitations, etc).
18. Not willing to avoid excessive sun exposure, steam baths, sauna, swimming and other strenuous activities during the study to ensure good scarring.
19. Not willing to refrain from use of skin care products applied on application sites for at least 5 days prior to start of Visit 2.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2014-01; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
AUC | during 12-36h of OFM-Sampling (post-dose)
  Area under the dOFM acyclovir concentration curve (AUC) during 12/36h of OFM-Sampling (post-dose)
CMAX | during 12-36h of OFM-Sampling (post-dose)
  Maximum observed dOFM acyclovir concentration (CMAX) during 12/36h of OFM-Sampling (post-dose)

SECONDARY OUTCOMES:
dOFM acyclovir concentration | during 12-36h of OFM-Sampling (post-dose)
TMAX | during 12-36h of OFM-Sampling (post-dose)
  Time to reach maximum dOFM acyclovir concentration (TMAX)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R Pieber, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University Graz, Graz, Styria, Austria